CLINICAL TRIAL: NCT04844879
Title: Prospective, Multicentre, Single-arm, Open, Confirmatory Trial to Assess Efficacy and Safety of a Navigation System Providing Personalized Soft Tissue Balance Data in Medially-stabilized Total Knee Arthroplasty
Brief Title: Medacta NextAR TKA Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02.022.02
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Diseases
Keywords: total knee arthroplasty; surgical navigation; medially-stabilized TKA
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): Patients suitable to receive Medacta GMK® Sphere system for primary TKA will be invited to take part to the study during the preoperative visit. Follow-ups are performed after 2, 6 and 12 months. Data collection includes clinical and radiological data for preoperative and postoperative assessments, as well as intraoperative details.
  Interventions: Device: NextAR TKA system

INTERVENTIONS:
Device: NextAR TKA system — The NextAR TKA system is a surgical guidance system which measures intra-operatively the effect of prosthesis alignment and positioning on soft tissue balance.

SUMMARY:
The goal of this study is to assess the efficacy and safety of a navigation system providing personalized soft tissue balance data in medially-stabilized total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
This is a prospective, multicentre, single-arm, open, confirmatory clinical investigation to assess the efficacy and safety of a navigation system providing personalized soft tissue balance data in medially-stabilized total knee arthroplasty (TKA).

Participants will be informed about the study, both orally and in writing, during a preoperative visit. The investigator will answer any questions that may arise and will collect the informed consent. During the study, enrolled participants will be able to withdraw at any time and for any reason.

The study is conducted according to the following schedule:

* V1 : Inclusion during a preoperative visit
* V2: Surgery
* V3: Follow-up visit at 2 month post-surgery
* V4: Follow-up visit at 6 months post-surgery
* V5: Follow-up visit at 12 months post-surgery

The following data will be collected:

* Oxford Knee Score (OKS), Knee Society Score (KSS), Forgotten Joint Score (FJS) and patient satisfaction at 6 months and 12 months of follow-up;
* Radiological analysis at 2 and 12 months of follow-up;
* Surgical time (min);
* Necessity of soft tissue release to obtain ligament or patellar balance;
* Time to discharge (days);
* Device deficiencies and peri- and postoperative adverse events.

A web-based data collection tool will be used as Electronic Data Capture (EDC). All the information required by the protocol will be collected in electronic case report forms (eCRF).

The statistical analysis will be performed according to a pre-established statistical analysis plan. Missing values will not be replaced by estimated values but will be considered as missing in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged over 18 years at time of surgery.
2. Patients who are scheduled to receive Medacta GMK® Sphere system for primary TKA (class III, CE-marked).
3. Patients with functional contralateral knee (i.e. without the need to use walking aids).
4. Patients willing and able to provide written informed consent for participation.
5. Patients willing to comply with the pre and post-operative evaluation schedule.

Exclusion Criteria:

1. Patients with one or more medical conditions identified as a contraindication defined by the labelling on any Medacta implants used in this study:

   * Patients presenting with progressive local or systemic infection
   * Muscular loss, neuromuscular disease or vascular deficiency of the affected limb, making the operation unjustifiable.
   * Severe instability secondary to advanced destruction of condralar structures or loss of integrity of the medial or lateral ligament
2. Patients whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems.
3. Patients affected by concomitant spine, hip, ankle or contralateral knee pathologies that can affect walking capacity.
4. Patients unable to understand and take action.
5. Patients with known allergy to the materials used.
6. Patients in which Medacta GMK® Sphere system is used in emergency interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Fucentese, Prof. Dr. med., Principal Investigator — Balgrist University Hospital
Locations (4):
- Switzerland (4):
  - Privatklinik Belair, Schaffhausen
  - Privatklinik Lindberg, Winterthur
  - Kantonsspital Winterthur, Winterthur
  - Uniklinik Balgrist, Zurich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Knees
Groups:
- NextAR TKA: Patients undergoing primary TKA with use of the navigation system providing personalized soft tissue balance data (Each unit represents a single patient)
Period: Overall Study
Arm/Group | NextAR TKA
Started | 40; 40 Knees (Each unit represents a single patient)
2-month Follow up | 40; 40 Knees
6-month Follow up | 39; 39 Knees
12-month Follow up | 37; 37 Knees
Completed | 37; 37 Knees
Not Completed | 3; 3 Knees
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- NextAR TKA: Patients undergoing primary TKA with use of the navigation system providing personalized soft tissue balance data
Arm/Group | NextAR TKA
Number analyzed (Participants) | 40
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 70.0 [51 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Oxford Knee Score [Median (Inter-Quartile Range); unit: score on a scale] — Range: 0-48; higher values indicate better outcomes
  score on a scale | 26.5 [20.0 to 29.0]
Forgotten Joint Score [Median (Inter-Quartile Range); unit: score on a scale] — Range: 0-100; higher values indicate better outcomes
  score on a scale | 15.6 [7.8 to 27.6]
Objective Knee Society Score [Median (Inter-Quartile Range); unit: score on a scale] — Range: 0-100; higher values indicate better outcomes.
  score on a scale | 45.5 [39.8 to 55.0]

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score (OKS)
Description: Oxford Knee Score (OKS) [Range: 0-48; higher values indicate better outcomes]
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | NextAR TKA
Number analyzed (Participants) | 39
scores on a scale | 39 [33 to 43]

2. Secondary Outcome: Oxford Knee Score (OKS)
Description: Oxford Knee Score (OKS) [Range: 0-48; higher values indicate better outcomes]
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | NextAR TKA
Number analyzed (Participants) | 37
score on a scale | 41 [36 to 46]

3. Secondary Outcome: Forgotten Joint Score (FJS)
Description: Forgotten Joint Score (FJS) [Range: 0-100; higher values indicate better outcomes]
Time Frame: 6 months and 12 months
Population: Lost at 6-month follow up: 1 Lost at 12-month follow up: 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | NextAR TKA
Number analyzed (Participants) | 39
score on a scale
  6-month follow up | 56.2 [30.2 to 78.1]
  12-month follow up: number analyzed (Participants) | 37
  12-month follow up | 60.4 [45.8 to 91.7]

4. Secondary Outcome: Objective Knee Society Score (KSS)
Description: Objective Knee Society Score (KSS) [Range: 0-100; higher values indicate better outcomes; total score reported as the average of subscale scores]
Time Frame: 6 months and 12 months
Population: Objective KSS. Lost at 6-month follow up: 1. Lost at 12-month follow up: 2.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | NextAR TKA
Number analyzed (Participants) | 39
score on a scale
  6-month follow up | 87.0 [63.0 to 96.0]
  12-month follow up: number analyzed (Participants) | 37
  12-month follow up | 88.5 [44.0 to 99.0]

5. Secondary Outcome: Radiological Outcomes
Description: X-ray assessment for the evaluation of: implant positioning, presence of radiolucent lines, subsidence, migration of components, presence of heterotopic ossifications or osteolysis
Time Frame: 2 months and 12 months
Population: Lost at 12-month follow up: 3
Measure: Count of Participants; unit: Participants
Arm/Group | NextAR TKA
Number analyzed (Participants) | 40
Participants
  2-month follow up: No Radiolucency (>2mm), Subsidence, Loosening | 40
  2-month follow up: Radiolucency (>2mm) - One Gruen Zone | 0
  2-month follow up: Subsidence | 0
  2-month follow up: Loosening | 0
  12-month follow up: number analyzed (Participants) | 37
  12-month follow up: No Radiolucency (>2mm), Subsidence, Loosening | 34
  12-month follow up: Radiolucency (>2mm) - One Gruen Zone | 3
  12-month follow up: Subsidence | 0
  12-month follow up: Loosening | 0

6. Secondary Outcome: Surgical Outcome - Surgical Time
Description: Surgical time (min)
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | NextAR TKA
Number analyzed (Participants) | 40
Participants
  60-80 minutes | 3
  81-100 minutes | 18
  101-120 minutes | 13
  121-150 minutes | 6

7. Secondary Outcome: Surgical Outcome - Necessity of Soft Tissue Release
Description: Necessity of soft tissue release to obtain ligament or patellar balance (Y/N)
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | NextAR TKA
Number analyzed (Participants) | 40
Participants | 0

8. Secondary Outcome: Surgical Outcome -Time to Discharge
Description: Time to discharge (days)
Time Frame: 2 months
Measure: Mean (Full Range); unit: days
Arm/Group | NextAR TKA
Number analyzed (Participants) | 40
days | 4.8 [3 to 16]

9. Secondary Outcome: Safety Outcomes
Description: Device deficiencies and adverse events
Time Frame: Intraoperative, 2 months, 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From signature of the informed consent up to 12 months postoperatively.
Description: All Serious adverse events are reported. Adverse events with at least "Unknown/Possible" relation with the procedure and/or the device are reported if rate exceeds 2.5%
Arm/Group | NextAR TKA
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 12/40
Other Adverse Events (participants affected / at risk) | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NextAR TKA (N=40)
Venous thrombosis (Blood and lymphatic system disorders) | 1 (1)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis flare (Musculoskeletal and connective tissue disorders) | 1 (1)
Accidental fall leading to TKA revision (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombosis main vein of the eye (Eye disorders) | 1 (1)
Accidental fall leading to wound opening and spine surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (General disorders) | 1 (1)
Transient deficit in range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic dislocation of the patella (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign paroxysmal positional vertigo (Ear and labyrinth disorders) | 1 (1)
Arthrosis contralateral knee (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NextAR TKA (N=40)
Postoperative knee pain, inflammation, or swelling (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT04844879/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT04844879/SAP_001.pdf